CLINICAL TRIAL: NCT03087227
Title: Evaluation of a Shared Health Information System for Home-hospital Management of Febrile NEUTROpenia After Cytotoxic Chemotherapy
Brief Title: Shared Health Information System for Febrile Neutropenia
Acronym: NEUTROSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marie-Helene METZGER (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor-Investigator, Marie-Helene METZGER, Dr, University of Paris 13
Organization: University of Paris 13 (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-009
Record Dates: First submitted 2017-02-20; First posted 2017-03-22 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Febrile Neutropenia; Solid Tumor; Hematologic Neoplasms
Keywords: mHealth; febrile neutropenia; neutropenia/chemically induced/*complications; antineoplastic agents/*adverse events; Patient readmission; disease management
MeSH Terms: conditions — Febrile Neutropenia; Hematologic Neoplasms; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEUTROSIS Intervention Group (Experimental): The NEUTROSIS Intervention group captures daily its temperature and the occurrence of other symptoms on the smartphone application. This information is then transmitted instantly to the hospital care team through the NEUTROSIS shared information system. The medical oncologist will be alerted in case of fever and will contact the patient.
  Interventions: Device: NEUTROSIS
- CONTROL Group (No Intervention): The control group will monitor daily its temperature and the occurrence of other symptoms on a paper surveillance diary and will have to contact the health team in case of fever as done in the usual care.

INTERVENTIONS:
Device: NEUTROSIS — evaluate a shared health information system (NEUTROSIS) for home-hospital management of febrile neutropenia after anti-tumor chemotherapy
  Arms: NEUTROSIS Intervention Group

SUMMARY:
The use of e-health in improving the quality of health services is a rapidly expanding research area, in particular its usefulness in patient management of the home-hospital care pathway. Febrile neutropenia is a serious and frequent complication of cytotoxic chemotherapy and better identification of low-risk patients who can be treated at home could be made possible by these technologies.

The objective of this study is to evaluate a shared health information system (NEUTROSIS) for home-hospital management of febrile neutropenia after anti-tumor chemotherapy. The study aims to compare the average length of hospital stay for febrile neutropenia among patients receiving NEUTROSIS and those receiving standard care

Materials and methods A shared information system (NEUTROSIS) has been developed to connect a smartphone web application for the patient to the existing shared medical record of the Paris Sud hospital group (AP-HP, France - 4D software).

The study consists of conducting a randomized controlled trial to compare a cohort of patients receiving cytotoxic chemotherapy for solid cancer or heamatological malignancies using the NEUTROSIS shared information system (n=100) and a cohort of patients followed by the hospital's standard care over a treatment period of six months (n=100). During the 15 days following each chemotherapy cycle, the 2 groups of patients must take their temperature daily. Both groups are trained like any patient under chemotherapy to contact the team in case of fever. The NEUTROSIS group captures daily its temperature and the occurrence of other symptoms on the smartphone application. This information is then transmitted instantly to the hospital care team who will be alerted in case of fever and will contact the patient. The control group will indicate these same data in a paper diary and will have to contact the health team in case of fever as done in the usual care.

The two groups of patients will be followed 6 months through a questionnaire asked to the patient at each hospital visit for chemotherapy cycle. The questionnaire collects information on the occurrence of symptoms and healthcare use between two chemotherapy cycles. A last follow-up questionnaire is asked by phone at the endpoint follow-up (6 months). The study will take place in two hospital sites of the Paris University hospital (A Béclère and Kremlin-Bicètre).

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Patient receiving cytotoxic chemotherapy for solid tumor or hematological malignancy
* Patient having signed consent to participate in the study
* Patient able to understand the protocol of care
* Patient covered by health insurance
* Patient with the use of a smartphone or tablet with Internet connection

Exclusion Criteria:

* patient refusing to participate in the study
* patient participating in a drug trial
* patient receiving or shifting to a weekly chemotherapy protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2019-10-20 (Actual)

PRIMARY OUTCOMES:
average length of hospital stay for febrile neutropenia | 6 months
  average length of hospital stay for febrile neutropenia

SECONDARY OUTCOMES:
hospitalisation rate | 6 months
  hospitalisation rate
healthcare use rate | 6 months
  emergency department, general practitioner,
Use rate | 6 months
  patient use rate

CONTACTS AND LOCATIONS:
Overall Officials: Francois BOUE, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hôpital Antoine Béclère, Clamart
  - Hôpital d'instruction des Armées de Percy, Clamart
  - Hôpital BICETRE, Le Kremlin-Bicêtre

IPD SHARING:
Plan to Share IPD: No